CLINICAL TRIAL: NCT00969033
Title: A Phase 2 Open-label Randomized, Controlled Trial of CS-1008 in Combination With Irinotecan Versus Irinotecan Alone in Subjects With Metastatic Colorectal Carcinoma Who Failed First-line Oxaliplatin Based Regimen
Brief Title: CS-1008 Used With Irinotecan Versus Irinotecan Alone in Subjects With Metastatic Colorectal Carcinoma Who Failed First-line Treatment With Oxaliplatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1008-A-E203
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tigatuzumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS-1008 with irinotecan (Experimental): CS-1008 and irinotecan
  Interventions: Drug: CS-1008; Drug: irinotecan
- irintoecan (Active Comparator): irinotecan alone
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: CS-1008 — CS-1008
  Arms: CS-1008 with irinotecan
Drug: irinotecan — irinotecan
  Other Names: Camptosar

SUMMARY:
The purpose of this study is to determine the effect of CS-1008 in combination with irinotecan compared to irinotecan alone on Progression-Free Survival (PFS) in subjects with metastatic or advanced colorectal cancer (CRC) who have failed oxaliplatin-based first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CRC which is now metastatic and after failure of oxaliplatin-based first-line treatment.
* At least 18 years of age.
* ECOG performance status =< 1.
* Measurable disease based on RECIST criteria.
* Adequate organ and bone marrow function as evidenced by:

  * Hemoglobin >= 9.0 g/dL (may be transfused to this level)
  * Absolute neutrophil count (ANC) >= 1.5 x 109/L
  * Platelet count >= 100 x 109/L
  * Serum creatinine =< upper limit of normal (ULN) or creatinine clearance > 50 mL/min
  * AST <= 2.5 x ULN in subjects with no liver metastasis and <= 5.0 x ULN in subjects with liver metastasis
  * Total bilirubin < 1.5 x ULN
* Men and women of childbearing potential must be willing to consent to using effective contraception (e.g., hormonal contraceptives, bilateral tubal ligation, barrier with spermicide, intrauterine device) while on treatment and for 3 months thereafter.
* All female subjects of childbearing potential must have a negative pregnancy test (serum or urine) result within 7 days before initiating study treatment.
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IEC/IRB approved ICF before performance of any study specific procedures or tests.
* Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Anticipation of need for a major surgical procedure or radiotherapy (RT) during the study.
* Treatment with chemotherapy hormonal therapy, RT, minor surgery, or any investigational agent within 4 weeks before study enrollment. Treatment with nitrosoureas, mitomycin C, immunotherapy, biological therapy, or major surgery within six weeks prior to study enrollment. St John's Wort within 2 weeks prior to study enrollment or during the study.
* History of any of the following conditions within 6 months before study enrollment:

  * Clinically significant myocardial infarction or severe/unstable angina pectoris
  * New York Heart Association (NYHA) class III or IV congestive heart failure (Section 17.2)
  * Clinically significant cerebrovascular accident, transient ischemic attack or pulmonary embolism- Clinically significant pulmonary disease (e.g., severe chronic obstructive pulmonary disease or asthma)
* Presence of any of the following: Symptomatic brain metastasis; an uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis.
* Clinically significant active infection that requires antibiotic therapy or Human Immunodeficiency Virus (HIV) positive subjects receiving antiretroviral therapy.
* History of malignancy other than CRC, unless there is the expectation that the malignancy has been cured, and tumor specific treatment for the malignancy has not been administered within the previous 5 years. Exceptions to this are non melanotic cancer of the skin and adequately treated carcinoma of the cervix-in-situ.
* Previous treatment with CS 1008, other agonistic DR5 antibody agents, or TRAIL agents.
* History of active chronic inflammatory bowel disease and/or bowel obstruction within the last 3 months.
* Pregnant or breast feeding.
* Known history of hypersensitivity reactions to irinotecan or to one of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine the difference in progression-free survival (PFS) for CS-1008 administered in combination with irinotecan and irinotecan alone. | 1 year

SECONDARY OUTCOMES:
Determine the difference in overall survival for CS-1008 administered in combination with irinotecan and irinotecan alone. | 1 year
Determine the difference in median survival for CS-1008 administered in combination with irinotecan and irinotecan alone. | 1 year
Determine the difference in objective response rate (ORR) for CS-1008 administered in combination with irinotecan and irinotecan alone. | 1 year
To determine the Incidence of anti- CS-1008 antibody formation. | 1 year

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Broomfield Hospital, Chelmsford, Essex
  - Mount Vernon Hospital, Northwood, Middlesex
  - Nottingham City Hospital, Nottingham, Notts
  - Chrichill Hospital, Oxford, Oxon
  - Royal Marsden Hospital, Sutton, Surrey
  - Clatterbridge Hospital, Bebington, Wirral
  - Royal United Hospital Bath, Bath
  - Russels Hall Hospital, Dudley
  - Leicester Royal Infirmary, Leicester